CLINICAL TRIAL: NCT05843981
Title: The Use of an Innovative, Thickened and Lasting Implant Comparing KS Versus TS Implants for Prosthetic Rehabilitations
Brief Title: Comparison KS Versus TS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Collaborators: Melodia, Dario, M.D. (Individual); Pisano, Milena, M.D. (Individual); Dr. Aurea Lumbau (Unknown); Prof. Silvio Mario Meloni (Unknown); Prof. Edoardo Baldoni (Unknown)
Responsible Party: Principal Investigator, Marco Tallarico, Assistant professor, Università degli Studi di Sassari
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNISS_PHD_Osstem_1
Record Dates: First submitted 2023-04-24; First posted 2023-05-06 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Dental Implant; Dental Implant-Abutment Design
Keywords: Dental Implant-Abutment Design; KS dental implant; Implant-abutment connection

STUDY DESIGN:
Intervention Model Description: Split-mouth
Who Masked: Participant, Outcomes Assessor
Masking Description: The patients, the outcome assessors (when possible) and the statistical advisors will be blind to the used implant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ks dental implant (Experimental): Innovative dental implant with lasting, internal conical connection of 15° and strengthened implant walls.
  Interventions: Device: Implant placement ks
- TSIII dental implant (Active Comparator): Standard dental implant with internal conical connection of 11°.
  Interventions: Device: Implant placement TS III

INTERVENTIONS:
Device: Implant placement TS III — Implant placement in subjects who have lost at least two teeth and need a prosthetic implant rehabilitation with TSIII Implant. . After osseointegration, dental implants will receive definitive prosthesis.
  Other Names: Dental prosthesis delivery
  Arms: TSIII dental implant
Device: Implant placement ks — Implant placement in subjects who have lost at least two teeth and need a prosthetic implant rehabilitation with KS Implant. After osseointegration, dental implants will receive definitive prosthesis.
  Other Names: Dental prosthesis delivery
  Arms: Ks dental implant

SUMMARY:
To compare the clinical and radiographic outcomes of two different implant systems with different implant-abutment connection: Osstem TS III (control group) versus Osstem KS (study group).

ELIGIBILITY:
Inclusion Criteria:

Any partially edentulous patient with partial edentulism, requiring at least two dental implant-supported rehabilitations, being 18 years or older, and able to sign an informed consent. Implant sites must allow the placement of two implants of at least 4 (premolars) or 4.5 (molars) mm of diameter and 8.5 mm of length. Smokers will be included and categorized into: 1) non smokers; 2) moderate smokers (smoking up to 10 cigarettes/day); 3) heavy smokers (smoking more than 11 cigarettes/day). In case of post-extractive sites, they must have been healing for at least 3 months before being treated in the study. Implants can be adjacent.

Exclusion Criteria:

* General contraindications to implant surgery.
* Patients irradiated in the head and neck area.
* Immunosuppressed or immunocompromised patients.
* Patients treated or under treatment with intravenous amino-bisphosphonates.
* Patients with untreated periodontitis.
* Patients with poor oral hygiene and motivation.
* Previous guided bone reconstruction at the intended implant sites.
* Uncontrolled diabetes.
* Pregnancy or nursing.
* Substance abuser.
* Psychiatric problems or unrealistic expectations.
* Lack of opposite occluding dentition in the area intended for implant placement.
* Patients with infection and or inflammation in the area intended for implant placement.
* Patients participating in other studies, if the present protocol cannot be properly adhered to.
* Patients referred only for implant placement and cannot be followed ant the treating centre.
* Patients unable to be followed for 5 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with implant failure | Up to 5 years
  Defined as implant mobility and/or any infection dictating implant removal, and/or implant fracture and/or any other mechanical complication rendering the implant unusable. The stability of each individual implant will be measured by the local blinded outcome assessors manually tightening the screws with a torque of 30 Ncm at abutment connection at initial loading. At 1,3 and 5 years after loading, individual implants will be manually tested for stability. Once the single crowns will be screwed, their stability will be assessed by rocking the crown with the handles of two dental instruments.
Number of Participants with prosthesis failure | Up to 5 years
  Whether it will not be possible to place the prosthesis because of implant failure or a prosthesis that has to be remade for any reason.
Number of complications | Up to 5 years
  Technical (fracture of the framework and/or the veneering material, screw loosening, etc.) and/or biologic (pain, swelling, suppuration, peri-implantitis, etc.) complications will be considered.

SECONDARY OUTCOMES:
Rate of peri-implant marginal bone level changes | At 1,3 and 5 years
  Peri-implant marginal bone level changes will be assessed on periapical radiographs took with the paralleling technique at implant placement, at initial loading, 1,3 and 5 years after loading. Ideally digital radiographs should be taken, otherwise radiographs on conventional films will be scanned into TIFF format with a 600 dpi resolution, and stored in a personal computer. Peri-implant marginal bone levels will be measured using the Scion Image (Scion Corporation, Frederick, MD, USA) software. The software will be calibrated for every single image using the known distance of the first two consecutive threads. Measurements of the mesial and distal bone crest level adjacent to each implant will be made to the nearest 0.01 mm. Reference points for the linear measurements will be: the coronal margin of the implant collar and the most coronal point of bone-to-implant contact. Bone levels will be measured.
Valuation of patient satisfaction | At 1,3 and 5 years
  Patients will answer the following questions (separately for each implant):
  1. Are you satisfied with the function of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  2. Are you satisfied with the aesthetic outcome of your implant-supported prostheses? Possible answers: yes absolutely, yes partly, not sure, not really, absolutely not.
  3. Would you undergo the same therapy again? Possible answers: "yes" or "no".

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tallarico, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No